CLINICAL TRIAL: NCT07338019
Title: The Buzdar Technique for Pulmonary Parenchymal Chest Tube Removal: Prospective Evaluation of a Novel Minimally Invasive Protocol
Brief Title: The Buzdar Technique
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Health Sciences Lahore (Other)
Responsible Party: Principal Investigator, Zeeshan Sarwar, Doctor, University of Health Sciences Lahore
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB/2025/1718/SIMS
Record Dates: First submitted 2026-01-03; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Chest Tube Management; Chest Tube Withdrawal; Iatrogenic Injury
Keywords: Pulmonary parenchymal chest tube (PPcT); chest tube malposition; tube thoracostomy complication; Buzdar technique; staged withdrawal

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pulmonary Parenchymal Tube Group (Experimental): The Buzdar Technique is a standardized, three-stage, minimally invasive approach designed to safely remove intraparenchymal chest tubes without thoracotomy or VATS. It aims to promote controlled fibrosis and gradual parenchymal healing before complete tube withdrawal.
  Interventions: Procedure: Gradual chest tube removal

INTERVENTIONS:
Procedure: Gradual chest tube removal — Stage 1: Healing and Fibrosis Phase (2 Weeks) Once PPcT is identified, the tube is left in situ for approximately 14 days to allow localized fibrosis and sealing of the injured lung parenchyma around the tube.
  During this period, the patient is kept under clinical observation and radiologic monitoring (serial chest X-rays or CT scan).
  Antibiotic coverage is continued to prevent secondary infection, and negative pressure drainage (closed chest drainage system) is maintained to ensure pleural space healing.
  Stage 2: Initial Retraction and Assessment After the initial 14-day period, under sterile conditions, the chest tube is retracted approximately 2 cm.
  If any resistance is encountered, gentle 360° rotation of the tube is performed to free adhesions.
  The patient is then observed for 24 hours, during which vital signs, oxygen saturation, and drainage output are monitored.
  A post-retraction chest X-ray is obtained to evaluate for pneumothorax, air leak, or any evidence of lung compromise

SUMMARY:
Chest tube thoracostomy remains a lifesaving intervention in trauma and thoracic surgery, used for the management of pneumothorax, hemothorax, empyema, and pleural effusions. Despite being one of the most frequently performed procedures worldwide, complication rates remain high, ranging from 20% to 40% [1]. Among these, pulmonary parenchymal chest tube (PPcT) insertion represents a rare but potentially devastating event, leading to hemorrhage, air leak, bronchopleural fistula, or infection. In Pakistan, where chest trauma and pneumothorax constitute major thoracic morbidities, PPcT cases are encountered with increasing frequency but remain underreported. Current literature describes only invasive surgical approaches-such as thoracotomy or video-assisted thoracic surgery (VATS)-for PPcT removal [9,10], with no established minimally invasive alternatives.

In response to this clinical challenge, the Department of Thoracic Surgery at (Hospital Name), Punjab, Pakistan, has developed and implemented a novel, minimally invasive three-stage removal technique, termed the Buzdar Technique, designed to ensure safe extraction of intraparenchymal chest tubes without surgical intervention. The technique follows a standardized protocol involving:

Healing phase: Tube left in situ for approximately two weeks to allow localized fibrosis and stabilization of the lung parenchyma.

Initial retraction: Gradual 2-cm withdrawal with optional 360° rotation under radiologic and clinical supervision, followed by 24-hour observation and chest imaging.

Sequential retractions: Weekly staged retractions of 2 cm until the last fenestration exits the pleural cavity, enabling safe final removal.

This prospective cohort study, conducted from July 2025 to June 2026, aims to evaluate the safety, effectiveness, and clinical outcomes of the Buzdar Technique in managing iatrogenic PPcT. Data will include patient demographics, procedural details, complications, radiologic recovery, and overall outcomes. Success will be defined as complete tube removal without pneumothorax, air leak, bleeding, or need for surgical intervention.

Preliminary institutional experience over the past decade has shown excellent results, with minimal morbidity, no requirement for thoracotomy or VATS, and full radiologic recovery in the majority of patients. The expected outcomes of this prospective evaluation are to validate these findings, establish the Buzdar Technique as a reproducible, evidence-based approach, and contribute to the global literature on non-surgical management of PPcT.

If proven effective, this technique could represent a paradigm shift in the management of intraparenchymal chest tubes-offering a safe, staged, and minimally invasive alternative to surgical removal, particularly beneficial for centers in low- and middle-income countries where advanced surgical options may not always be available.

DETAILED DESCRIPTION:
Chest tube thoracostomy remains a cornerstone in the management of pleural and thoracic pathologies, including pneumothorax, hemothorax, empyema, and pleural effusions. By lowering intrapleural pressure and promoting lung re-expansion, it ensures adequate tissue oxygenation and effective ventilation [1, 2]. Despite its widespread use, complication rates following tube thoracostomy remain high-ranging from 20% to 40%-and include insertional, positional, and infectious events. Pneumothorax and chest trauma are among the major causes of thoracic morbidity in Pakistan. In a Karachi-based study, 40% of 146 pneumothorax cases were attributed to traumatic and iatrogenic causes, with intercostal tube drainage utilized in 81% of patients. Similarly, another study reported that 35% of thoracic trauma patients experienced tube-related complications such as empyema and bronchopleural fistula. These findings underscore the urgent need for procedural standardization, improved operator training, and enhanced complication management strategies.

Tube thoracostomy is a frequently performed procedure in emergency and trauma care settings, taught in most surgical and medical training curricula and standardized within the Advanced Trauma Life Support (ATLS) program. Nevertheless, globally, insertion-related complications continue to present significant clinical challenges. International literature has emphasized the importance of standardized classification and reporting systems for chest tube-related complications, broadly categorizing them into insertional, positional, removal, infectious, and device-related events. The implementation of such standardized systems and adherence to best-practice protocols have been shown to reduce complication rates significantly-from 12.6% to as low as 4.4% in some trauma centers.

Among insertional complications, pulmonary parenchymal chest tube (PPcT) represents one of the most serious, occurring when the chest tube inadvertently traverses into the lung tissue. PPcT is particularly associated with patients who have pleural adhesions, poor pulmonary compliance, or consolidated lungs. Despite its potential to cause catastrophic outcomes such as bleeding or bronchopleural fistula, PPcT remains underreported and lacks standardized management guidelines. Reported interventions for removal are limited to invasive surgical approaches such as thoracotomy with thoracoplasty and video-assisted thoracic surgery (VATS) without lung resection. However, no literature currently describes minimally invasive, staged, or gradual removal techniques for such cases.

At the Department of Thoracic Surgery, Services Hospital, Lahore, Punjab, Pakistan, several cases of PPcT have been managed over the last decade. In response to this clinical challenge, our team developed a novel, minimally invasive three-stage removal strategy, termed the Buzdar Technique, initiated in 2006. This standardized protocol aims to achieve safe removal of intraparenchymal chest tubes without the need for thoracotomy or VATS while minimizing morbidity and preventing recurrence or pneumothorax. The method involves: (1) leaving the tube in situ for approximately two weeks to promote localized fibrosis; (2) gradual 2-cm retractions with optional 360° rotation under radiologic and clinical monitoring, followed by a 24-hour observation and chest radiograph; and (3) sequential weekly retractions until the last fenestration exits the pleural space, at which point safe removal is achieved.

This prospective cohort study, conducted from July 2025 to June 2026, aims to evaluate the effectiveness, safety, and clinical outcomes of the Buzdar Technique for managing pulmonary parenchymal chest tubes. By documenting its results systematically, this study seeks to provide evidence for a reproducible, less invasive alternative to surgical extraction, potentially establishing a new standard of care in managing PPcT.

Objectives:

* To evaluate the effectiveness and safety of the Buzdar Technique for the removal of pulmonary parenchymal chest tubes (PPcT) in patients managed at a tertiary thoracic surgery center.
* To assess the clinical outcomes, including complication rates (bleeding, air leak, pneumothorax, empyema) and duration of hospital stay following application of the technique.
* To determine the radiological and functional recovery of lung parenchyma after staged removal using the Buzdar Technique.
* To establish this method as a standardized minimally invasive approach for the management of iatrogenic PPcT cases.

Hypothesis:

The Buzdar Technique, a minimally invasive three-stage removal protocol for pulmonary parenchymal chest tubes, is a safe, effective, and reproducible method that minimizes morbidity, prevents complications, and eliminates the need for surgical interventions such as thoracotomy or video-assisted thoracoscopic surgery (VATS).

Methods and Materials

Study Design and Duration:

This will be a prospective cohort study conducted in the Department of Thoracic Surgery, Services Hospital, Lahore, Punjab, Pakistan, over two years (July 2025 - June 2027). All eligible patients with iatrogenic pulmonary parenchymal chest tube (PPcT) insertion confirmed by radiological evidence will be enrolled after informed consent.

Sample Size and Selection:

Sample Size: All the patients that are expected to meet the inclusion criteria during the study period.

Inclusion Criteria:

* Patients ≥18 years with confirmed intraparenchymal chest tube placement on chest CT or X-ray.
* Hemodynamically stable patients suitable for conservative staged removal.
* Patients providing informed consent.

Exclusion Criteria:

* Patients requiring immediate thoracotomy due to massive bleeding or large bronchopleural fistula.
* Patients with uncorrectable coagulopathy or unstable cardiopulmonary status.
* Patients refusing participation or lost to follow-up.

Data Collection Parameters:

Data will be prospectively recorded using a standardized proforma and include:

* Demographics: age, gender, comorbidities.
* Etiology: trauma, iatrogenic, or post-procedural causes.
* Radiological Findings: tube position, depth of parenchymal penetration, associated lung injury.
* Procedural Data: duration from insertion to initiation of Buzdar Technique, total number of retraction stages, total duration of tube in situ.
* Outcomes: incidence of air leak, pneumothorax, bleeding, infection, duration of hospital stay, need for surgical intervention, and radiologic resolution.

Description of the Buzdar Technique:

The Buzdar Technique is a standardized, three-stage, minimally invasive approach designed to safely remove intraparenchymal chest tubes without thoracotomy or VATS. It aims to promote controlled fibrosis and gradual parenchymal healing before complete tube withdrawal.

Stage 1: Healing and Fibrosis Phase (2 Weeks) Once PPcT is identified, the tube is left in situ for approximately 14 days to allow localized fibrosis and sealing of the injured lung parenchyma around the tube.

During this period, the patient is kept under clinical observation and radiologic monitoring (serial chest X-rays or CT scan).

Antibiotic coverage is continued to prevent secondary infection, and negative pressure drainage (closed chest drainage system) is maintained to ensure pleural space healing.

Stage 2: Initial Retraction and Assessment After the initial 14-day period, under sterile conditions, the chest tube is retracted approximately 2 cm.

If any resistance is encountered, gentle 360° rotation of the tube is performed to free adhesions.

The patient is then observed for 24 hours, during which vital signs, oxygen saturation, and drainage output are monitored.

A post-retraction chest X-ray is obtained to evaluate for pneumothorax, air leak, or any evidence of lung compromise.

Stage 3: Sequential Retractions and Final Removal Weekly retractions of approximately 2 cm are continued under radiologic and clinical supervision until the last fenestration of the chest tube exits the pleural cavity.

At each stage, the patient undergoes 24-hour monitoring and radiological assessment before proceeding further.

When the tube's last side hole lies outside the pleural space and the lung remains expanded, the tube is removed completely under controlled conditions.

A final chest radiograph is performed to confirm complete lung expansion and absence of pneumothorax.

Throughout the process, no general anesthesia or surgical intervention is required, and patients are typically managed on an inpatient basis or under short-stay observation. The staged, fibrosis-based approach minimizes the risk of parenchymal tearing, air leak, or hemorrhage, which are common during abrupt tube extraction.

Outcome Measures:

Primary Outcome: Successful removal of the PPcT without pneumothorax, significant air leak, or bleeding.

Secondary Outcomes: Duration of hospitalization, rate of infection or empyema, radiologic lung re-expansion, and need for further surgical intervention.

Statistical Analysis:

Data will be analyzed using SPSS version 26.0. Continuous variables will be presented as mean ± standard deviation, while categorical variables will be expressed as percentages and frequencies. The success rate of the technique and complication incidence will be calculated. Associations between demographic and clinical factors and outcomes will be assessed using the Chi-square test or Fisher's exact test, with a p-value <0.05 considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥18 years with confirmed intraparenchymal chest tube placement on chest CT or X-ray.
* Hemodynamically stable patients suitable for conservative staged removal.
* Patients providing informed consent.

Exclusion Criteria:

* Patients requiring immediate thoracotomy due to massive bleeding or large bronchopleural fistula.
* Patients with uncorrectable coagulopathy or unstable cardiopulmonary status.
* Patients refusing participation or lost to follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Complete chest tube removal | 02 weeks
  Successful removal of the Pulmonary Parenchymal chest Tube without pneumothorax, significant air leak, or bleeding.

CONTACTS AND LOCATIONS:
Locations (1):
- Services Hospital Lahore, Lahore, Punjab Province, Pakistan